CLINICAL TRIAL: NCT00898443
Title: Success Rate, Efficiency, and Predictors of Reactivation of a Continuous Labor Epidural Catheter for Postpartum Tubal Ligation
Brief Title: Continuous Labor Epidural Catheter for Tubal Ligation Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Marsha Wakefield, MD, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: F080829007
Record Dates: First submitted 2009-05-08; First posted 2009-05-12 (Estimated); Results first posted 2012-08-07 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-06

CONDITIONS: Tubal Ligation; Bilateral Tubal Ligation
MeSH Terms: interventions — Anesthesia, Spinal

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Spinal Anesthetic Group (Other): This group will receive spinal anesthetic for the surgical procedure and will serve as the control group for this study.
  Interventions: Other: Spinal anesthetic
- Epidural Anesthetic Group (Experimental): This is the experimental group for this study.
  Interventions: Other: Epidural anesthetic

INTERVENTIONS:
Other: Epidural anesthetic — Use of the existing continuous labor epidural for surgical anesthetic for postpartum tubal ligation
  Arms: Epidural Anesthetic Group
Other: Spinal anesthetic — This group was assigned to receive spinal anesthetic for postpartum tubal ligation.
  Arms: Spinal Anesthetic Group

SUMMARY:
This study is to study the success rate of using the epidural catheter that was placed during the labor for the surgical anesthesia to perform a postpartum tubal ligation.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) 1-3 postpartum women desiring Postpartum Bilateral Tubal Ligation (PPBTL) for infertility
* Functional epidural catheter placed for labor and delivery analgesia
* The epidural is still taped within 1cm of the original depth when it was functional for labor analgesia
* 1-45 years of age

Exclusion Criteria:

* ASA 4 status
* History of dural puncture ("wet tap") during initial epidural catheter insertion
* History of marginal or inadequate epidural analgesia for labor
* Cesarean section for delivery
* Examination demonstrates that the indwelling catheter has migrated more than 1 cm from the original depth when secured
* The end of indwelling epidural catheter appears to have not been capped appropriately or the cap was not maintained intact
* Prolonged sensory or motor block, bladder or anal sphincter dysfunction, nerve damage, inability to ambulate, post-dural puncture headache (PDHD), or seizures, during or after delivery and following cessation of the epidural catheter dosing
* Pseudocholinesterase deficiency
* Allergy to Nesacaine® (chloroprocaine) or lidocaine
* General anesthesia provided for delivery
* History of substance abuse disorder
* History of major psychiatric disorder
* Non-English reading/speaking participants

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2008-10; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marsha L. Wakefield, MD, Principal Investigator — UAB Department of Anesthesiology
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women in labor, admitted to UAB Labor & Delivery, who requested postpartum tubal ligation after delivery.
Period: Overall Study
Arm/Group | Spinal Anesthetic Group | Epidural Anesthetic Group
Started | 10 | 8
Completed | 9 | 8
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Spinal Anesthetic Group | Epidural Anesthetic Group | Total
Number analyzed (Participants) | 9 | 8 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 8 | 17
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 8 | 17

OUTCOME MEASURES:

1. Primary Outcome: Success Rate of Reactivation of Existing Continuous Labor Epidural Catheter for Postpartum Tubal Ligation
Description: Rate of reactivation of the epidural catheter for postpartum tubal ligation in the group that was randomized to the epidural anesthetic group. (Need for additional supplemental analgesics and sedatives or the need to convert to general anesthesia.)
Time Frame: at the time of surgery
Population: Only the patients who were recruited, randomized and had all their data completed at the time of their procedure were included in the analysis. Insufficient numbers were recruited to complete the study as designed.
Measure: Number; unit: participants
Arm/Group | Spinal Anesthetic Group | Epidural Anesthetic Group
Number analyzed (Participants) | 9 | 8
participants | 0 (0) | 7 (0)

2. Secondary Outcome: Impact of Anesthesia Type on OR (Operating Room) Efficiency
Description: The time minutes)from initiation of anesthesia to surgery start.
Time Frame: minutes until surgery start
Population: as for outcome 1
Measure: Median (Full Range); unit: minutes
Arm/Group | Spinal Anesthetic Group | Epidural Anesthetic Group
Number analyzed (Participants) | 9 | 8
minutes | 14 [8 to 22] | 29 [19 to 37]

ADVERSE EVENTS:
Time Frame: 48 hours after procedure
Description: If the subject was discharged before they were seen by the research nurse, an attempt was made to call them within 48 hours.
Arm/Group | Spinal Anesthetic Group | Epidural Anesthetic Group
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/8
Other Adverse Events (participants affected / at risk) | 0/9 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes